CLINICAL TRIAL: NCT05385692
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of Injectable BL-M02D1 in Patients With Locally Advanced or Metastatic Gastrointestinal Tumors or Other Solid Tumors
Brief Title: A Study of BL-M02D1 in Patients With Locally Advanced or Metastatic Gastrointestinal Tumors or Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M02D1-102
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Digestive Tract Tumors; Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M02D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M02D1

INTERVENTIONS:
Drug: BL-M02D1 — Administration by intravenous infusion

SUMMARY:
In phase Ia study, the safety and tolerability of BL-M02D1 in patients with locally advanced or metastatic gastroenteric tumor or other solid tumors will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) of BL-M02D1.

In phase Ib study, the safety and tolerability of BL-M02D1 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

In addition, the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-M02D1 in patients with locally advanced or metastatic gastroenteric tumor or other solid tumors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must sign the informed consent form voluntarily and follow the plan requirements.
2. No gender limit.
3. Age: ≥18 years old and ≤75 years old (phase Ia); ≥18 years old (phase Ib).
4. Expected survival time ≥ 3 months.
5. Locally advanced or metastatic gastrointestinal tumor and other solid tumor confirmed by histopathology and/or cytology, which are incurable or currently without standard treatment.
6. Agree to provide archived tumor tissue samples or fresh tissue samples from the primary tumor or metastatic tumor within 2 years (TROP2 protein expression in tumor pathological tissue to explore the correlation between TROP2 protein expression and bl-M02D1 validity index); If subjects are unable to provide tumor tissue samples, they will be admitted after evaluation by the investigator if other admission criteria are met.
7. Participants must have at least one measurable lesion that meets the definition of RECIST v1.1 in phase Ib.
8. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
9. Toxicity of previous antitumor therapy has returned to ≤ level 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic laboratory abnormalities considered by the investigators, such as elevated ALP, hyperuricemia, and elevated blood glucose; Toxicities with no safety risk were excluded, such as alopecia, hyperpigmentation, and grade 2 peripheral neurotoxicity. Or decreased hemoglobin except ≥90 g/L).
10. Has adequate organ function before registration, defined as: a) Bone marrow function: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet count ≥90×109/L, Hemoglobin ≥90 g/L; B) Hepatic function: Total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN for participants without liver metastasis, AST and ALT ≤5.0 ULN for liver metastases; c) Renal function: Creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to the Cockcroft and Gault formula).
11. Coagulation function: International normalized ratio (INR)≤1.5×ULN, and activated partial thromboplastin time (APTT)≤1.5ULN.
12. Urinary protein ≤2+ or ≤1000mg/24h.
13. For premenopausal women with childbearing potential, a pregnancy test must be taken within 7 days prior to the start of treatment. Serum or urine pregnancy must be negative and must be non-lactating. Adequate barrier contraceptive measures should be taken during the treatment and 6 months after the end of treatment for all participants (regardless of male or female).

Exclusion Criteria:

Patients screened for any of the following conditions will not be included in this study:

1. Antitumor therapy such as chemotherapy, biotherapy, immunotherapy, radical radiotherapy, major surgery (as defined by the investigators), and targeted therapy (including small-molecule tyrosine kinase inhibitors) within 4 weeks prior to initial administration or within 5 half-lives, whichever is shorter; Mitomycin and nitrosourea were administered within 6 weeks before the first administration; Oral fluorouracil drugs such as Tizio, capecitabine, or palliative radiotherapy within 2 weeks before first administration; Traditional Chinese medicines with anti-tumor indications were administered within 2 weeks before the first dose.
2. Prior treatment with ADC drugs targeting TROP2 or ADC drugs using camptothecin derivatives (topoisomerase I inhibitors) as toxins.
3. Participants with history of severe heart disease, such as: symptomatic congestive heart failure (CHF) ≥ grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ grade 2 heart failure, history of transmural myocardial infarction, unstable angina pectoris, Left ventricular ejection fraction < 50% etc.
4. Participants with prolonged QT interval (male QTc> 450 msec or female QTc> 470 msec), complete left bundle branch block, III grade atrioventricular block.
5. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for type I diabetes, hypothyroidism that can be controlled only by alternative treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis).
6. The presence of a second primary tumor within 5 years prior to initial administration, except for radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resected carcinoma in situ.
7. Screening for unstable thrombotic events such as deep vein thrombosis, arterial thrombosis and pulmonary embolism requiring therapeutic intervention within the first 6 months; Infusion device-related thrombosis is excluded;
8. Patients with poorly controlled pleural effusion with clinical symptoms were judged by researchers to be unsuitable for inclusion.
9. Participants with poorly controlled hypertension by antihypertensive drugs (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg).
10. Lung disease defined as grade ≥3 according to CTCAE V5.0; ≥2 grade of radioactive lung disease, current or history of interstitial lung disease (ILD).
11. Symptoms of active central nervous system metastasis. However, participants with stable brain metastasis can be included. Stable is defined as: a. With or without antiepileptic drugs, the seizure-free state lasts for more than 12 weeks; b. There is no need to use glucocorticoids; c. Continuous multiple MRI (scanning interval at least 8 weeks) showed a stable state in imaging; d. Stable after treatment for more than 1 month without symptoms;
12. Participants who have a history of allergies to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-M02D1.
13. Participants have a history of organ transplantation or allogeneic stem cell transplantation (Allo-HSCT).
14. In the adjuvant (or neoadjuvant) treatment of anthracyclines, the cumulative dose of anthracyclines is> 360 mg/m2.
15. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number> the lower limit of detection) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > the lower limit of detection).
16. Participants with active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
17. Participated in another clinical trial within 4 weeks prior to participating in the study.
18. Pregnant or nursing women.
19. Other conditions that the investigator believes that it is not suitable for participating in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M02D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M02D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M02D1.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-M02D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M02D1 will be investigated.
T1/2 | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M02D1 will be investigated.
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to 21 days after the first dose
  CL in the serum of BL-M02D1 per unit of time will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-M02D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of BL-M02D1 will be evaluated.
Nab (neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of BL-M02D1 will be evaluated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M02D1 to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China